CLINICAL TRIAL: NCT03009955
Title: Comparison of Postoperative Pain Between Patients Received Primary and Repeated Caesarean Section
Status: Completed | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Hong Li, Director, Department of Anesthesiology, Xinqiao Hospital of Chongqing
Other Study IDs: Postoperative pain
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Caesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group P: patients who received primary caesarean section
- Group R: patients who received repeated caesarean section

SUMMARY:
To everyone knows, more and more patients received repeated caesarean section in China. However, at present it is not known what is it like about their postoperative pain intensity, and is it different from those patients who received primary caesarean section. Thus through postoperative follow-up, the current study aimed to investigate and compare the postoperative pain between patients received primary and repeated caesarean section.

DETAILED DESCRIPTION:
According to whether or not to receive repeated caesarean patients were grouped into group P or group R. For all maternal,standardized epidural anesthesia and caesarean section were performed. Then the pain VAS scores and Ramsay scores at 4h, 8h, 12h, 24h and 48h after the surgery were recorded. And sleep quality at 1 day and 2 day after the surgery were recorded. In addition, pain situation at 1 week and 4 weeks after the surgery was followed up.

ELIGIBILITY:
Inclusion Criteria:

* single birth
* full-term pregnancy
* in accordance with cesarean section indications
* transverse incision of lower uterine segment

Exclusion Criteria:

* history of dementia, psychiatric illness or any diseases of central nervous system
* accompanying liver or kidney function deficiency
* alcoholism and drug dependence
* patients previously included in this study or currently included in the other clinical study
* patients who have second surgery during the study period
* difficult to follow up or patients with poor compliance
* history of chronic pain

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who receiving primary and repeated caesarean section.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2016-12; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain VAS at 4, 8, 12, 24 and 48 hours after the surgery | At 4, 8, 12, 24 and 48 hours after the surgery

SECONDARY OUTCOMES:
Pain intensity at 3 to 7 days after the surgery | At 3 to 7 days after the surgery
Pain intensity at 4 weeks after the surgery | At 4 weeks after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Li, M.D., Principal Investigator — Department of Anesthesiology, Xinqiao Hospital, Third Military Medical University
Locations (1):
- Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duan G, Yang G, Peng J, Duan Z, Li J, Tang X, Li H. Comparison of postoperative pain between patients who underwent primary and repeated cesarean section: a prospective cohort study. BMC Anesthesiol. 2019 Oct 22;19(1):189. doi: 10.1186/s12871-019-0865-9. PMID 31640565